CLINICAL TRIAL: NCT02571621
Title: Evaluation of Serial Usage of Combitube in Anesthesiology
Brief Title: Serial Usage of Combitube in Anesthesiology
Acronym: Combitube
Status: Completed | Type: Observational
Sponsor: Michael Frass (Other)
Responsible Party: Sponsor-Investigator, Michael Frass, Professor, Medical Doctor, Medical University of Vienna
Organization: Medical University of Vienna (Other)
Other Study IDs: 2015/10
Record Dates: First submitted 2015-10-01; First posted 2015-10-08 (Estimated); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Surgery

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients intubated with Combitube: Patients with Combitube intubation undergoing general anesthesia with ASA class I and II
  Interventions: Device: Combitube

INTERVENTIONS:
Device: Combitube — Intubation with Combitube

SUMMARY:
Retrospective evaluation of a database of ETC routine uses during general anaesthesia.

DETAILED DESCRIPTION:
Background: The oesophageal-tracheal Combitube (ETC) was designed for the use in the pre-hospital setting and has proven its value both there and in difficult airway management. The ETC is a double-lumen tube and as such it enables ventilation independent of its position in either the trachea or the oesophagus. Since laryngoscopy is not necessary for positioning the ETC, it is especially favoured in pre-hospital setting, but is also used in clinical setting.

Objectives: Retrospective evaluation of a database of ETC routine uses during general anaesthesia.

ELIGIBILITY:
Inclusion Criteria:

* patients ASA class I and II

Exclusion Criteria:

* patients not able to sign informed consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients undergoing general anesthesia physical status ASA class I and II
Sampling Method: Non-Probability Sample
Enrollment: 745 (Actual)
Dates: Start 1989-01; Primary Completion 2006-06 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Success rate | 3 minutes
  Measurement time in seconds using a stopwatch between grasping the tube and successful intubation

SECONDARY OUTCOMES:
BMI | 1hour
  Measurement of Body mass index by calculating height and weight of each patient
method of insertion and size of the tube, | 1hour
  insertion with different intubation devices and diameters of tubes
Intubator's qualification and experience in the use of the ETC; | 1 hour
  years of training and experience in intubators as well as use of ETC for at least 10 times

CONTACTS AND LOCATIONS:
Overall Officials: Michael Frass, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Med. Univ. Vienna, Dept. Internal Med. I, Vienna, Austria

REFERENCES:
- [Result] Sethi AK, Desai M, Tyagi A, Kumar S. Comparison of combitube, easy tube and tracheal tube for general anesthesia. J Anaesthesiol Clin Pharmacol. 2014 Oct;30(4):526-32. doi: 10.4103/0970-9185.142849. PMID 25425779